CLINICAL TRIAL: NCT01026415
Title: An Open-Label Clinical Pharmacology Study of Brentuximab Vedotin (SGN-35) in Patients With CD30-Positive Hematologic Malignancies: CYP3A4 Drug-Drug Interactions, Excretion, and Special Populations
Brief Title: Clinical Pharmacology Study of Brentuximab Vedotin (SGN-35)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-008
Expanded Access: NCT01196208 (No longer available)
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Carcinomas; Disease, Hodgkin; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin; Neoplasms
Keywords: Antibody-Drug Conjugate; Antigens, CD30; Disease, Hodgkin; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin; monomethyl auristatin E; Drug Therapy; Immunotherapy; Hematologic Diseases; Lymphoma; Antibodies, Monoclonal
MeSH Terms: conditions — Carcinoma; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin; Neoplasms; Hematologic Diseases; Lymphoma | interventions — Brentuximab Vedotin; Rifampin; Midazolam; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): midazolam +/- brentuximab vedotin
  Interventions: Drug: brentuximab vedotin; Drug: midazolam
- 2 (Experimental): brentuximab vedotin +/- rifampin
  Interventions: Drug: brentuximab vedotin; Drug: rifampin
- 3 (Experimental): brentuximab vedotin +/- ketoconazole
  Interventions: Drug: ketoconazole; Drug: brentuximab vedotin
- 4 (Experimental): special populations
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg IV every 21 days
  Other Names: ADCETRIS; SGN-35
  Arms: 1; 2
Drug: rifampin — 600 mg/day PO
  Arms: 2
Drug: midazolam — 1 mg IV
  Arms: 1
Drug: ketoconazole — 400 mg/day PO
  Arms: 3
Drug: brentuximab vedotin — 1.2 mg/kg IV every 21 days
  Other Names: SGN-35
  Arms: 3; 4

SUMMARY:
The purpose of this study is to identify brentuximab vedotin drug-drug interactions in patients with CD30-positive cancers and to determine the main route of excretion. The study will also assess blood drug levels in patients with renal or hepatic impairment (special populations).

ELIGIBILITY:
Inclusion Criteria:

* Adequate organ function (Special Populations: serum bilirubin >2 mg/dL or creatinine clearance <50 mL/min)
* ECOG performance status <2 (Special Populations: <4)
* Relapsed or refractory CD30-positive malignancy

Exclusion Criteria:

* Receiving prohibited medication within 4 weeks
* Poor liver function (Child-Pugh class C)
* Current diagnosis of primary cutaneous ALCL
* Acute or chronic graft-versus-host disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Midazolam blood concentrations +/- brentuximab vedotin | 3 weeks
Brentuximab vedotin blood concentrations +/- rifampin | 6 weeks
Brentuximab vedotin in urine, feces, and blood | 1 week
Brentuximab vedotin blood concentrations in special populations | 3 weeks
Brentuximab vedotin blood concentrations +/- ketoconazole | 6 weeks

SECONDARY OUTCOMES:
Incidence of adverse events and laboratory abnormalities | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Manley, MD, Study Director — Seagen Inc.
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - St. Francis Medical Group Oncology & Hematology Specialists, Indianapolis, Indiana
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Seattle Cancer Care Alliance / University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Result] Han TH, Gopal AK, Ramchandren R, Goy A, Chen R, Matous JV, Cooper M, Grove LE, Alley SC, Lynch CM, O'Connor OA. CYP3A-mediated drug-drug interaction potential and excretion of brentuximab vedotin, an antibody-drug conjugate, in patients with CD30-positive hematologic malignancies. J Clin Pharmacol. 2013 Aug;53(8):866-77. doi: 10.1002/jcph.116. Epub 2013 Jun 10. PMID 23754575
- [Derived] Gopal AK, Ramchandren R, O'Connor OA, Berryman RB, Advani RH, Chen R, Smith SE, Cooper M, Rothe A, Matous JV, Grove LE, Zain J. Safety and efficacy of brentuximab vedotin for Hodgkin lymphoma recurring after allogeneic stem cell transplantation. Blood. 2012 Jul 19;120(3):560-8. doi: 10.1182/blood-2011-12-397893. Epub 2012 Apr 17. PMID 22510871